CLINICAL TRIAL: NCT01316796
Title: A Phase I Study of the Use of Topical Sodium Nitrite for Chronic Leg Ulcers in Adult Patients With Hemolytic Disorders
Brief Title: Topical Sodium Nitrite for Chronic Leg Ulcers in Adult Patients With Blood Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110121; 11-H-0121
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10-12

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease; Chronic Hemolytic Disorders
Keywords: Sickle Cell Disease; Hemolysis; Anemia; Nitric Oxide; Blood Flow; Leg Ulcer; Sickle Cell Anemia; Thalassemia; Hemolytic Blood Disorder
MeSH Terms: conditions — Anemia, Sickle Cell; Hemolysis; Anemia; Leg Ulcer; Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Sodium Nitrite Cream

SUMMARY:
Background:

- Chronic leg ulcers are a complication of many blood disorders such as sickle cell disease, thalassemia, and other red blood cell disorders. In these disorders, red blood cells break down earlier than normal, which researchers suspect may cause or contribute to the development of leg ulcers; however, the exact cause is unknown, and current therapies are not very effective. Researchers are interested in determining if a research cream made with sodium nitrite, a substance that is known to increase blood flow by dilating blood vessels, may speed up the healing of skin ulcers.

Objectives:

- To evaluate the safety and effectiveness of topical sodium nitrite cream as a treatment for chronic leg ulcers in individuals with sickle cell disease or other red blood cell disorders.

Eligibility:

- Individuals at least 18 years of age who have sickle cell disease or another red cell disorder and have had a leg ulcer for more than 4 weeks.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and an examination of the ulcer, including x-ray of the leg(s) with the ulcer and swabs from the wound.
* Participants will be scheduled for a 5-day inpatient stay at the Clinical Center, with the following procedures:
* Days 1 and 2: Participants will have blood draws, a wound assessment, ultrasound of the affected leg, imaging studies (magnetic resonance imaging and infrared photography), thermo-patch application to monitor temperature changes, measurements of blood flow in the skin, and questionnaires about pain and quality of life. An optional skin biopsy may also be conducted with samples taken near the skin ulcer
* Day 3: Participants will have one ulcer treated with the topical cream. Frequent blood draws will be conducted before application and then regularly for up to 6 hours after application of the cream. Thirty minutes after the research cream is applied, participants will have imaging studies of the treated leg and measurements of pain levels and blood flow.
* Day 4: Participants will have a blood draw and temperature recordings taken.
* Day 5: Participants will have the research cream applied and the same imaging studies as before, and will be discharged for care at home.
* For the following 3 weeks, participants will come to the clinical center twice a week to have the research cream applied to the leg ulcer and tests performed by the study researchers.
* For the fourth and final week, participants will return for additional cream treatment sessions, imaging studies, blood draws, and other tests as directed by the study researchers.
* Study participation will end in the following week (week 5). Subjects will come for a final visit one month after the end of the study.

DETAILED DESCRIPTION:
Leg ulcerations have long been identified as a serious and debilitating complication of SCD and even the first SCD patient described in North America in 1910 had leg ulcerations. The prevalence varies, being low before 10 years of age, and in genotypes other than SS, and it is influenced by geographical location, with an occurrence as high as 75 percent of SS patients in Jamaica, and 8-10 percent in North America. The etiology of chronic ulcers in SCD and other hemolytic disorders is unknown, mechanical obstruction by dense sickled red cell, increased venous pressure, bacterial infections, abnormal autonomic control with excessive vasoconstriction when in the dependent position, degree of anemia with decrease in oxygen carrying capacity, and in situ thrombosis, have all been proposed as potential contributing factors. Recent studies have reported increased incidence of leg ulcers in patients with pulmonary hypertension. Our group has pioneered the notion of an association between the hemolytic phenotype and leg ulcers. Current treatment options for leg ulcerations, including antibiotics, compression bandages, dressing changes, Unna boots, silver and zinc oxide gauze, skin grafts and maggot therapy rely mostly on bacterial containment, stimulation of granulation formation and decrease of venostasis. Pathological changes in the microcirculation associated with ulceration are not addressed. Nitric oxide metabolism has been the focus of our branch research over the past several years. We know that it mediates essential biological processes, including vasodilatation, wound healing, and angiogenesis and has antimicrobial activity. Moreover, NO has an antiplatelet effect and influences several growth factors involved in endothelial homeostasis.

We propose a Phase I study of a topical cream containing escalating doses of sodium nitrite, a local donor of NO when in the presence of heme, as a novel approach to the therapy for chronic leg ulcers in hemolytic disorders. The primary objectives are to evaluate topical sodium nitrite cream s safety and tolerability in patients with sickle cell disease or other hemolytic disorders and chronic leg ulcers and to determine the optimal concentration of the study drug that is tolerated. Subjects will be treated at the Clinical Center for 4 weeks.

Potential benefit will be a durable resolution or improvement of the leg ulcer. Possible side effects include hypotension and methemoglobinemia, secondary to sodium nitrite absorption for the ulcerated skin. Safety measures will be used and pharmacokinetics analysis of sodium nitrite absorption in this setting will be obtained. As a secondary endpoint, we will study the biology of leg ulcer formation in patients with hemolytic disorders, its pathological appearance on a skin biopsy, and the role of microvascular changes in its formation and (possibly) resolution. Sophisticated and novel studies of blood flow and temperature changes during sodium nitrite application, as well as macrovascular appearance on MRI will allow for a better understanding of ulcer formation. This may lead to novel approaches to the therapy of ulcer in hemolytic and non-hemolytic disorders, such as diabetes and decubitus ulceration.

ELIGIBILITY:
* INCLUSION CRITERIA:

Each subject must meet all of the following inclusion criteria during the screening process in order to participate in the study:

* Subjects must have a diagnosis of sickle cell disease (SS, SC, S-beta-thalassemia), other hemoglobinopathies, or hemolytic disorders, such as hereditary spherocytosis.
* Be at least 18 years old.
* Have a leg ulcer of at least 4 weeks (28 days) duration.
* Leg ulcer must be no smaller than 2.5 cm(2) and no larger than 100 cm(2).
* Provide written informed consent.

EXCLUSION CRITERIA:

Subjects meeting any of the following criteria during baseline evaluation will be excluded from entry into the study:

* Exposure to therapeutic nitric oxide, L-arginine, nitroprusside or nitroglycerine within the past 1 week.
* Subjects presenting with clinically diagnosed bacterial infection (e.g., osteomyelitis, pneumonia, sepsis or meningitis).
* Subjects who have a pre-existing methemoglobinemia (more than 2.5 percent), unless the cytochrome b5 reductase (methemoglobin reductase) is within normal limits and the methemoglobin is no greater than 3 percent)
* Patients who are currently enrolled in any other investigational drug study (this does not include observational or natural history protocols).
* Use of PDE5 inhibitors, such as sildenafil, 4 days prior to screening.
* Pregnant women (urine or serum HCG plus) or nursing mothers.
* The following list of drugs and agents may cause methemoglobinemia and should be avoided while on this study:

  * Anesthetics (local): Benzocaine, procaine, prilocaine, Anbesol, Orajel
  * Antimalarials: chloroquine, primaquine, quinacrine
  * Aniline dyes
  * Chlorates
  * Dapsone
  * Diarylsulfonylureas
  * Doxorubicin
  * Metoclopramide
  * Nitric and nitrous oxide
  * Nitrobenzenes (shoe and floor polish and in paint solvents)
  * Nitroethane (artificial nail remover, propellent, fuel additive)
  * Nitrofurantoin (furadantin)
  * Pyridium (phenazopyridine)
  * Phenacetin (acetaminophen)
  * Phenylhydrazine
  * Rasburicase
  * Sulfonamides (sulfacetamide, sulfamethoxazole, sulfanilamide, sulfapyridine)

    * If a subject participant meets exclusion criteria while participating in the trial, then the subject will be removed from the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03-15; Primary Completion 2015-09-18 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Evaluate topical sodium nitrite cream's safety and tolerability in patients with sickle cell disease or other hemolytic disorders and chronic leg ulcers.
Determine the optimal concentration of topical nitrite cream that is tolerated.

SECONDARY OUTCOMES:
Determine whether changes of local temperature correlates with ulcer appearance, modification, or healing.
Determine whether topical nitrite therapy changes regional blood flow to the affected skin area and surrounding.
Determine whether it shows preliminary evidence for accelerating wound healing.
Determine the pharmacokinetics of topical sodium nitrite cream and methemolglobin profile in patients with sickle cell disease.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Hsieh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Herrick JB. Peculiar elongated and sickle-shaped red blood corpuscles in a case of severe anemia. 1910. Yale J Biol Med. 2001 May-Jun;74(3):179-84. No abstract available. PMID 11501714
- [Background] Akinyanju O, Akinsete I. Leg ulceration in sickle cell disease in Nigeria. Trop Geogr Med. 1979 Mar;31(1):87-91. PMID 483376
- [Background] Koshy M, Entsuah R, Koranda A, Kraus AP, Johnson R, Bellvue R, Flournoy-Gill Z, Levy P. Leg ulcers in patients with sickle cell disease. Blood. 1989 Sep;74(4):1403-8. PMID 2475188
- [Derived] Minniti CP, Gorbach AM, Xu D, Hon YY, Delaney KM, Seidel M, Malik N, Peters-Lawrence M, Cantilena C, Nichols JS, Mendelsohn L, Conrey A, Grimes G, Kato GJ. Topical sodium nitrite for chronic leg ulcers in patients with sickle cell anaemia: a phase 1 dose-finding safety and tolerability trial. Lancet Haematol. 2014 Dec 1;1(3):e95-e103. doi: 10.1016/s2352-3026(14)00019-2. PMID 25938131